CLINICAL TRIAL: NCT05259306
Title: Low-Intensity Focused Ultrasound of the Mediodorsal Thalamus for Treatment-resistant Schizophrenia: Circuit Interrogation and Symptom Assessment
Brief Title: Low-Intensity Focused Ultrasound Neuromodulation of the Mediodorsal Thalamus for Treatment-Resistant Schizophrenia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Indefinite hold due to administrative issues.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-01291
Record Dates: First submitted 2022-01-18; First posted 2022-02-28 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Treatment-resistant Schizophrenia
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment-resistant Schizophrenia group (Experimental): The subject will present for three baseline visits, followed by a treatment visit and subsequently follow-up visits at 24-hours, 48-hours, 1 week, 2 weeks, 1 month, and 3 months. Feasibility will be assessed as well as symptoms via detailed symptom rating scales at each visit. At the treatment visit itself, participants will undergo MR-guided low-intensity focused ultrasound of the MD thalamus.
  Interventions: Device: Insightec Exablate Neuro MR-guided focused ultrasound transducer

INTERVENTIONS:
Device: Insightec Exablate Neuro MR-guided focused ultrasound transducer — This study will be utilizing the Insightec Exablate Neuro MR-guided focused ultrasound transducer to deliver low-intensity ultrasonic energy precisely and safely to the target region of the brain. MRgFUS has been FDA approved at high-intensity to treat essential tremor and Parkinson's disease associated tremor. Device premarket approval number (PMA) is P150038, and FDA approval notice was July 11, 2016. This study will be using this device not to make any lesions in the brain (as it is currently FDA approved), but instead to use the precision and non-invasive nature of the device to target the MD thalamus region of the brain at intensities currently approved by the FDA for transcranial ultrasound.

SUMMARY:
This pilot study aims to investigate the use of MRI-guided low-intensity focused ultrasound (LIFU) to modulate neuronal activity within the thalamus in human subjects with treatment-resistant schizophrenia.

DETAILED DESCRIPTION:
Approximately 30% of patients with schizophrenia have symptoms that persist despite multiple antipsychotic medication trials including clozapine, and there is currently no evidence-based treatment option for this population. These patients often suffer psychological distress related to their psychotic symptoms, become chronically disabled, and are unable to lead meaningful lives. Several promising new treatment modalities are being explored including deep brain stimulation (DBS) in subjects with treatment-resistant schizophrenia. A pilot study at another institution is using DBS of the substantia nigra pars reticulata (SNr) to modulate circuitry in the thalamus by disinhibiting the mediodorsal (MD) nucleus of the thalamus. This approach follows evidence from multiple structural and functional studies implicating hypofunction of the MD thalamus in the pathophysiology of schizophrenia. This includes an association between MD hypofunction and both positive and cognitive symptoms of schizophrenia including auditory hallucinations and working memory, respectively. As DBS is an invasive neurosurgical procedure with small but definable risks of neurologic injury, a minimally invasive screening method to optimize patient selection for DBS would be optimal.

This pilot study aims to investigate the use of MRI-guided low-intensity focused ultrasound (LIFU) to modulate neuronal activity within the thalamus in human subjects with treatment-resistant schizophrenia. Focused ultrasound itself is a safe, incisionless technology with high spatial resolution and depth penetration that has been shown to stimulate and inhibit neuronal activity. At high intensities, focused ultrasound can be used to thermally ablate a specific region of brain tissue and has been FDA-approved for the treatment of essential tremor and tremor in Parkinson's disease via thermal ablation of the ventral intermediate (VIM) thalamus. In contrast, LIFU is non-ablative and thus can be used for transient neuromodulation with high spatial precision due to direct real-time MRI targeting. This pilot study aims to use non-ablative LIFU to target the MD thalamus noninvasively and specifically, with the aim of interrogating and modulating the neuronal circuitry involved in symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has an age greater or equal to 21 years old.
* Subject has a diagnosis of schizophrenia as determined by a review of medical records, discussion with referring psychiatrist, as well as the Structured Clinical Interview for DSM-5 (SCID-5).
* Subject is determined to be treatment-resistant for at least one year prior to Visit 1 as demonstrated by clinical evidence (determined via medical records and referring psychiatrist) of persistent auditory hallucinations and/or delusions that have not responded to treatment with three adequate trials/regimens of antipsychotic medication, as follows:

  a. Adequate trials of any two different antipsychotic medications, belonging to different classes of at least 12 weeks equivalent to at least 500 mg/day of chlorpromazine within the previous five years.
* Subject has a score of at least moderate (4) on two of the three BPRS positive symptoms (conceptual disorganization, hallucinatory behavior, and unusual thought content) at all three Baseline Visits.
* Subject must be ambulatory.
* Female subjects must be practicing an acceptable method of contraception, postmenopausal, physically incapable of childbearing, or; if practicing an acceptable method of contraception, a negative urine pregnancy test must be confirmed at all three Baseline Visits
* Subject has decision-making capacity to provide informed consent, as determined by an independent psychiatrist.

Exclusion Criteria:

* Subject has a positive urine toxicology screen at any of the three Baseline Visits.
* Subject has medical contraindications to the procedure as determined by an internist or primary care physician.
* Subject is pregnant or breast-feeding.
* Subject has a history of alcohol or substance abuse within the past 6 months.
* Subject has a medical illness, comorbid psychiatric illness, and/or abnormal diagnostic finding that would interfere with the completion of the study, confound the results of the study, or pose risk to the patient.
* Subject has participated in another investigational drug trial or therapeutic trial within 30 days of Baseline Visit 1.
* Subject has a neurologic condition or history of traumatic brain injury associated with loss of consciousness and/or intracranial bleeding.
* Subject is considered high suicide risk as screened by the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Subject has a defibrillator, pacemaker, or other implants that would interfere with MRI
* Subject has significant social factors that greatly interfere with consistent follow up and/or support.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of Patients who Complete All Visits Related to the Study | Up to Month 3
  Measurement of feasibility of low-intensity focused ultrasound (LIFU) for treatment-resistant schizophrenia. Feasibility defined as two out of three patients completing all visits related to the study.

SECONDARY OUTCOMES:
Change in Brief Psychiatric Rating Scale (BPRS) Score from Baseline | Baseline, Month 3
  BPRS is a measurement of the severity of schizophrenia. It assesses the level of 18 symptom constructs including hostility, suspiciousness, hallucination, and grandiosity. The rater enters a number for each symptom construct that ranges from 1 (not present) to 7 (extremely severe), while items that are not assessed are scored as 0. The total score is the sum of responses and ranges from 18 to 126; higher scores indicate greater severity of symptoms.
Change in Positive and Negative Syndrome Scale (PANSS) Score from Baseline | Baseline, Month 3
  PANSS is a 30-item medical scale used for measuring symptom severity of patients with schizophrenia. Items are rated on a 7-point scale (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, and 7=extreme). The total score is the sum of responses and ranges from 30 to 210; higher scores indicate greater illness severity.
Change in Montreal Cognitive Assessment (MoCA) Score from Baseline | Baseline, Month 3
  MoCA is a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total score is the sum of responses and ranges from 0 to 30; higher scores indicate less cognitive dysfunction. A normal score is defined as greater than or equal to 26.

CONTACTS AND LOCATIONS:
Overall Officials: Alon Mogliner, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Requests should be directed to alon.mogilner@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.